CLINICAL TRIAL: NCT06641765
Title: Continuous Glucose Monitoring in Haemodialysis and Peritoneal Dialysis Patients With Type 1 and Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring in Dialysis Patients With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Feldt-Rasmussen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, MD, DMSc, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGM-Dialysis study
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Continuous Glucose Monitoring; Haemodialysis; Peritoneal Dialysis
Keywords: Hypoglycaemia; Quality of life; Time-in-range; HbA1c; Diabetes; Dialysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomized controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control group (Group 1) (No Intervention): Will undergo standard glycaemic monitoring (HbA1c and finger-prick glucose) along with 10 days double-blinded CGM sessions scheduled at months 0, 3, 6, and 9.
  Glucose-lowering treatment is adjusted by an endocrinologist or a diabetes nurse at months 0, 3, and 6.
  CGM data will be double-blinded, and treatment adjustments will be based on usual monitoring of HbA1c and finger-prick glucose.
- Intermittent CGM (Group 2) (Active Comparator): Will have intermittent access to 10 days of open CGM scheduled at months 0, 3, 6 along with double-blinded CGM at month 9.
  Glucose-lowering treatment is adjusted by an endocrinologist or a diabetes nurse at months 0, 3, and 6.
  The objective is to adjust their glucose-lowering treatment to ensure patients spend less than 1% of their time with glucose levels below 3.9 mmol/L and more than 60% of the time within the target range (3.9 to 10.0 mmol/L).
  Interventions: Device: Continous Glucose Monitoring
- Continuous CGM (Group 3) (Active Comparator): Will have continuous access to open CGM throughout the entire duration of the study from month 0-9.
  Glucose-lowering treatment is adjusted by an endocrinologist or a diabetes nurse at months 0, 3, and 6.
  The objective is to adjust their glucose-lowering treatment to ensure patients spend less than 1% of their time with glucose levels below 3.9 mmol/L and more than 60% of the time within the target range (3.9 to 10.0 mmol/L).
  Interventions: Device: Continous Glucose Monitoring

INTERVENTIONS:
Device: Continous Glucose Monitoring — 10 days of real time open access to Continous Glucose Monitoring - either at defined time intervals (Group 2) or continuously for 9 months (Group 3).
  Other Names: Dexcom G7
  Arms: Continuous CGM (Group 3); Intermittent CGM (Group 2)

SUMMARY:
The primary objective of this multicenter, randomized controlled trial is to assess whether the intermittent or continuous use of continous glucose monitoring can enhance glycaemic control among dialysis patients with type 1 or type 2 diabetes, in comparison to the standard monitoring involving finger-prick glucose and HbA1c.

Participants will be monitored for 9 months and randomly assigned to one of three groups:

* Group 1, the control group, will undergo standard monitoring (using HbA1c and BGM) along with double-blinded CGM sessions at month 0, 3, 6, and 9.
* Group 2 will have intermittent access to open CGM during the same time intervals.
* Group 3 will have continuous access to open CGM throughout the entire duration of the study.

During the study period, participants will have three consultations with an endocrinologist for adjustments in their glucose-lowering treatment.

The goal is to compare markers of glycaemic control between the three groups. Secondary objectives include evaluating the impact on hypoglycaemia, quality of life, hospitals admissions and cardiovascular events.

DETAILED DESCRIPTION:
INTRODUCTION

Dialysis patients with diabetes have a very short life expectancy likely caused by a high incidence of co-morbidities combined with an increased risk of hypoglycaemia and poor glycaemic control. Glycaemic monitoring is a challenge in dialysis patients, and the number of available glucose-lowering agents are reduced often necessitating the use of insulin. Overall, this means that dialysis patients do not receive the same high quality of treatment as the general diabetes population.

In the past decades various diabetes technologies have revolutionised treatment, primarily in type 1 diabetes, but have also shown effect in type 2 diabetes. Continuous glucose monitoring (CGM) is a device applied to the skin that provides a detailed glucose profile which enables the endocrinologist to tailor and optimize diabetes treatment. We hypothesise that intermittent and/or continuous utilization of CGM will significantly improve glycaemic control for patients undergoing haemodialysis or peritoneal dialysis, thereby potentially reducing complications associated with diabetes in this population.

OBJECTIVES

The primary objective is to assess whether the intermittent or continuous use of CGM can enhance glycaemic control among dialysis patients with type 1 or type 2 diabetes, in comparison to the standard-monitoring involving finger-prick glucose and HbA1c.

Secondary objectives include assessing the impact of CGM on hypoglycaemia incidence, quality of life, and cardiovascular events.

BACKGROUND

The combination of diabetes and end-stage renal disease is associated with a high risk of diabetic complications with a mean survival time of 3 to 4 years. To reduce the risk of diabetic complications, glycaemic control is essential, where the aim is to avoid both hypo- and hyperglycaemia. For patients undergoing dialysis, HbA1c is currently the most widely used tool for glycaemic monitoring. However, several studies have found HbA1c to be an unreliable glycaemic marker. In addition, glycaemic targets using HbA1c are not provided in current guidelines as studies report conflicting results on the optimal HbA1c target. Therefore, new approaches for glycaemic control are warranted to improve diabetes treatment.

Continuous glucose monitoring (CGM):

CGM uses a subcutaneous sensor to measure glucose levels every 5 to 15 min depending on the model. A CGM provides a detailed estimate of the glucose profile and studies in patients with type 1 and type 2 diabetes have demonstrated that CGM-use improved glycaemic control without increasing the risk of hypoglycaemic events.

A CGM provides several glycaemic indexes including mean sensor glucose, variables for glucose variability, time-in-ranges and are used to adjust antidiabetic treatment. Time-in-ranges is a relatively new tool in glycaemic control where the percentage time spent in different glucose intervals is calculated from the measured CGM data, for a period (typically 10 to 14 days). Time-in-ranges are defined as the percentage time spent in time-below-range (<3.9 mmol/L); time-in-target-range (3.9 to 10.0 mmol/L); time-above-range (>10.0 mmol/L) mmol/L). The advantage of using time-in-ranges for glycaemic control is the ability to diminish the risk of hypoglycaemia while maintaining glycaemic control by optimizing the time spent in the target-range.

Current use of CGM in dialysis patients:

Two minor studies have used CGM to adjust the antidiabetic treatment in patients receiving dialysis. These studies reported that the use of CGM with subsequent adjustment in antidiabetic treatment was associated with a reduction in HbA1c level and could indicate a beneficial effect of CGMs in the dialysis population8. However, a CGM-based approach to diabetes treatment is not well defined and is currently bases on a consensus report recommending patients with high risk of hypoglycaemia (which includes dialysis patients) achieving the following glycaemic targets using time-in-ranges:

* More than 50% time within time-in-target-range (3.9-10.0 mmol/L) (>12 h per day)
* Less than 1% spent below-range (<3.9 mmol/L) (<15 min per day)
* Less than 50% above-range (>10.0 mmol/L) (<12 h per day)
* Less than 10% above 13.9 mmol/L (<2 h and 24 min per day) However, these recommendations have not been evaluated in dialysis patients and it remains unknown if these targets provide sufficient glycaemic control, reduce complications, improves quality of life or are practical feasible.

The technical aspects of daily CGM use could constitute a problem for some of the most fragile dialysis patients. Intermittent use of CGMs could therefore be an alternative approach and have, in non-dialysis patients with diabetes, lead to a lowering of elevated HbA1c levels. Intermittent CGM usage could alleviate the practical burden on both patients and medical staff, reduce expenses, and still equip endocrinologists with CGM data for optimizing glycaemic control. However, recent advancements in CGM technology have enhanced usability and continuous use of CGMs likely hold advantages over intermittent usage.

DESIGN AND POPULATION

This multicentre, prospective, randomized controlled study will be conducted at Rigshospitalet, Roskilde University Hospital, North Zealand Hospital Hillerød, Herlev Hospital, and Holbæk Hospital, encompassing all dialysis centres in eastern Denmark.

The study will include a total of 96 participants with type 1 or type 2 diabetes undergoing either haemodialysis or peritoneal dialysis. Participants will be randomly assigned in a 1:1:1 ratio to either receive standard glycaemic monitoring (Group 1), intermittent CGM (Group 2) or continuous CGM (Group 3).

METHODS

All participants will be monitored for 9 months and randomly assigned to one of three groups (Figure 3). Group 1, the control group, will undergo standard monitoring (using HbA1c and finger-prick glucose) along with double-blinded CGM sessions scheduled at months 0, 3, 6, and 9. Group 2 will have intermittent access to open CGM during the same time intervals. Meanwhile, Group 3 will have continuous access to open CGM throughout the entire duration of the study.

All three groups will undergo a 10-day period of double-blinded CGM to assess their baseline glucose profiles. Additionally, participants will have three consultations with an endocrinologist or a diabetes nurse at months 0, 3, and 6 for adjustments in their glucose-lowering treatment. At the final visit (month 9), Groups 1 and 2 will undergo a 10-day period of double-blinded CGM, while Group 3 will have an open CGM session.

The objective for the intervention groups (Group 2 and 3) is to adjust their glucose-lowering treatment to ensure patients spend less than 1% of their time with glucose levels below 3.9 mmol/L and more than 60% of the time within the target range (3.9 to 10.0 mmol/L). Meanwhile, for the control group, CGM data will be double-blinded, and adjustment of glucose lowering medicine will be based on usual monitoring of HbA1c and finger-prick glucose.

STATISTICAL ANALYSIS

Statistical analysis is performed as intention-to-treat and will be conducted by the investigators in close collaboration with an experienced statistician. All data will be described including data-incompleteness as well as reasons for data-incompleteness. A linear mixed model with a participant-specific random intercept is used to analyse the effect of changes in mean sensor glucose, time in range and HbA1c. This analysis will compare changes across the three study groups from baseline to end of the study.

ETHICAL CONSIDERATIONS

CGM is a well-tested technology that has significantly improved glucose management in the general diabetes population. It is expected to be safe and well tolerated, in dialysis patients as well. The many examinations are time consuming for the study participants. The project, however, will likely yield important knowledge on how to optimize diabetes management in dialysis patients, which expectedly will benefit both the study participants and in general all dialysis patients with diabetes.

The study will be registered at ClinicalTrials.gov prior to initiation. The trial protocol adheres to the principles of the Helsinki Declaration II, and the study will be conducted in compliance with Good Clinical Practice, the Act on the Processing of Personal Data, and the General Data Protection Regulation. Approval from the regional Research Ethical Committees are underway. Participants are covered by The Patient Compensation Association.

PERSPECTIVES

We expect that blood glucose regulation tailored to CGM, instead of HbA1c/finger prick will improve blood glucose levels and reduce the incidence of hypoglycemia among dialysis patients. We expect the project to contribute to rethinking diabetes treatment among these patients, leading to increased survival, reduced diabetes complications and hospitalizations, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial-related procedures are performed
* Diabetes, one of the following groups: Type 1 diabetes OR Type 2 diabetes receiving glucose-lowering therapy OR Type 2 diabetes managed with lifestyle changes with an HbA1c ≥ 50 mmol/mol
* Maintenance haemodialysis or peritoneal dialysis (minimum of two weeks)
* Subject must be willing and able to comply with trial protocol and be fluent in Danish or English

Exclusion Criteria:

* Major allergy to tape/adhesives
* Women who are pregnant or planning pregnancy
* Ongoing use of CGM
* Ongoing use of insulin pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in time-in-target-range (3.9-10 mmol/L) from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.

SECONDARY OUTCOMES:
Difference in percentage of participants reaching the goal of minimum of 60% of time-in-target-range (3.9-10 mmol/L) between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in time-in-range < 3 mmol/L from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in time-in-range < 3.9 mmol/L from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in time-in-range 3.9-7.8 mmol/L from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline ,months 0, 3, 6, and 9.
Change in time-in-range > 10 mmol/L from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in time-in-range > 13.9 mmol/L from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in Mean Sensor Glucose (mmol/L) from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in Glucose Variability (SD (mmol/L) and coefficient of variation (%)) from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in HbA1c (%, mmol/mol) from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Change in Glucose Management Indicator (%, mmol/mol) from baseline through to study end between the three groups. | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Difference in length of time-period with active CGM between the three groups | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Difference in incidence of CGM time in <3.0mmol/L range lasting >15 minutes between the three groups | 9 Months
  Evaluated by 10 days of CGM obtained at baseline, months 0, 3, 6, and 9.
Difference in incidence of severe hypoglycaemia (Requiring third party assistance) between the three groups | 9 Months
  Evaluated by medical records and patient interview at months 0, 3, 6, and 9.
Difference in incidence of Adverse Events (AE) and Adverse Device Events between the three groups | 9 Months
  Evaluated by medical records and patient interview at months 0, 3, 6, and 9.
Difference in incidence of Serious Adverse Events (SAE) and Serious Adverse Device Events between the three groups | 9 Months
  Evaluated by medical records and patient interview at months 0, 3, 6, and 9.
Difference in incidence of Suspected Unexpected Serious Adverse Reactions (SUSAR) between the three groups | 9 Months
  Evaluated by medical records and patient interview at months 0, 3, 6, and 9.

OTHER OUTCOMES:
Difference in "Hypoglycaemia Fear Survey [HFS-II]" between the three groups | 9 Months
  Evaluated by questionnaire "Hypoglycaemia Fear Survey [HFS-II]" at baseline and end of trial
Difference in "The Diabetes Treatment Satisfaction Questionnaire status" between the three groups | 9 Months
  Evaluated by questionnaire "The Diabetes Treatment Satisfaction Questionnaire status [DTSQs]" at baseline and the end of trial and "The Diabetes Treatment Satisfaction Questionnaire change [DTSQc]" at the end of trial.
Difference in "Gold Score" (Hypoglycaemia awareness) between the three groups | 9 Months
  Evaluated by questionnaire "Gold Score" at baseline and the end of trial
Difference in "Clarke Score" (Hypoglycaemia awareness) between the three groups | 9 Months
  Evaluated by questionnaire "Clarke Score" at baseline and the end of trial
Difference in "SARC-F questionnaire" (Frailty) between the three groups | 9 Months
  Evaluated by questionnaire "SARC-F" at baseline and the end of trial
Difference in "Problem Areas in Diabetes [PAID]" (Diabetes distress) between the three groups | 9 Months
  Evaluated by questionnaire "Problem Areas in Diabetes [PAID]" at baseline and the end of trial
Change in weight from baseline to study end between the three groups | 9 Months
  Measured at baseline and end of trial
Change in pulse (beats per minute) from baseline through to study end between the three groups | 9 Months
  Measured at baseline and months 3, 6, and 9 (measured twice with an automatic device using left or right arm after 10 min of sitting at rest).
Change in blood pressure (mmHg) from baseline through to study end between the three groups | 9 Months
  Measured at baseline and months 3, 6, and 9 (measured twice with an automatic device using left or right arm after 10 min of sitting at rest).
Difference in incidence cardiac events (arrhythmias and acute myocardial infarction) between the three groups | 9 Months
  Evaluated by review of medical records at baseline and months 3, 6, and 9.
Difference in number of days of hospitalization during the study period between the three groups | 9 Months
  Evaluated by review of medical records. Counted from months 3 to 9. (Additionally, the number of hospitalizations days in the 6 months preceding the baseline visit is counted to assess baseline equivalence between groups)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bomholt, MD, PhD, Principal Investigator — Department of Nephrology, Rigshospitalet, University of Copenhagen
Locations (5):
- Denmark (5):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - North Zealand Hospital, Hillerød, Hillerød
  - Holbæk Sygehus, Holbæk
  - Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No